CLINICAL TRIAL: NCT05272579
Title: PrePhage - Faecal Bacteriophage Transfer for Enhanced Gastrointestinal Tract Maturation in Preterm Infants - Clinical Trial
Brief Title: PrePhage - Faecal Bacteriophage Transfer for Enhanced Gastrointestinal Tract Maturation in Preterm Infants
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lise Aunsholt, Neonatologist, Clinical Professor (Unknown)
Responsible Party: Principal Investigator, Gustav Riemer Jakobsen, Medical Doctor, Ph.d-student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rigshospitalet - PrePhage
Record Dates: First submitted 2022-02-15; First posted 2022-03-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Necrotizing Enterocolitis; Microbial Substitution
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Intervention Model Description: In a block randomized trial with 14 days of follow up between each step, a total of 10 infants will be treated with fecal filtrate transfer and 10 infants will be treated with placebo. The structure will be: 2+2, 2+2, 2+2, 6+6
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFT treatment (Experimental): Treatment with fecal filtrate transfer in saline solution administered by nasogastric tube
  Interventions: Other: Fecal Filtrate Transfer
- Placebo Treatment (Placebo Comparator): Treatment with saline solution administered by nasogastric tube
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal Filtrate Transfer — Treatment with donated fecal samples filtered to contain practically no bacteria and mainly viruses, including bacteriophages
  Arms: FFT treatment
Other: Placebo — Saline solution
  Arms: Placebo Treatment

SUMMARY:
PrePhage - Fecal bacteriophage transfer for enhanced gastrointestinal tract maturation in preterm infants

This pilot triol has the primary goal of demonstrating the safety of transferring viruses and proteins from healthy term infants to preterm infants born between gestational age (GA) 26 + 0 and 30+6. The long-term goal is to develop a safe and effective treatment to prevent the severe gut disease called necrotizing enterocolitis (NEC).

NEC is a common disease in neonatal intensive care units affecting 5-10% of all admitted patients. 15-30% of the affected children die from the disease, and many of the survivors suffer from the effects of extensive gut surgery.

While the disease is caused by many different factors, recent research has shown the gut microbiome to be a central factor in the development of NEC. Furthermore, in the recent years special viruses called bacteriophages have shown potential in the treatment of various diseases.

By collecting feces from healthy, term infants and filtering it thoroughly, the investigators can provide a treatment that contains practically only viruses, proteins and nutrients. It is our belief that giving the preterm infants a mix of viruses including bacteriophages will prevent NEC.

To do this, the investigators will go through 3 stages:

1. Recruiting and following healthy donor infants to study the microbiota and use feces from them to donate in stage 2 and 3
2. Examining the safety of the treatment as well as how it works in preterm piglets
3. Testing the treatment in preterm infants. 10 preterm infants will receive the treatment and 10 preterm infants will receive placebo. The investigators expect to see no serious side effects to the treatment. The investigators hope, but do not expect to be able to see a beneficial effect of the treatment.

If this pilot trial shows promising results, it will be followed be a larger clinical trial.

DETAILED DESCRIPTION:
PrePhage - Fecal bacteriophage transfer for enhanced gastrointestinal tract maturation in preterm infants

This pilot trial aims to investigate if fecal filtrate transfers (FFT) to preterm infants is safe and tolerable. To investigate this, the investigators will recruit 20 donor infants and their mothers from time of delivery, and both will be subjected to a novel screening program including blood, urine, breastmilk, fecal screening and standard clinical investigation. Donor fecal samples will be collected from time of birth and with varying intervals for consecutive 3 years for 3 purposes: 1) to conduct safety studies in preterm piglets before transfer to preterm recipient infants, 2) to conduct FFT to preterm infants, and 3) to map normal microbiota development in healthy infants. The feces used for donation will be collected between 2-4 weeks after birth. After 1 year, donated feces will be released for FFT to preterm, but only if the donor infant at this time has been healthy and normally developed. Donors are followed up for consecutive 3 years after birth. Maternal fecal samples will be compared to infant samples, to investigate maternal to infant transfer of microbiota, as well as changes in infant microbiota in response to environment.

20 preterm infants with gestational age between 26 +0 - 30+6 weeks + days, are block randomized to either FFT or saline placebo within 24 hours after birth and the following 3 days, in total 4 donations. The recipients are clinically and biochemically closely monitored by attending staff and the group of investigators according to best clinical practice and predefined clinical observation. The recipients are followed up for consecutive 3 years to evaluate potential late side-effects and to monitor change in fecal microbiome after transplant or placebo.

The primary endpoint is to assess safety of FFT to preterm infants with expected no increase in necrotizing enterocolitis (NEC), sepsis and death in the intervention group. The secondary endpoint is to assess if, FFT treatment will reduce incidence of feeding tolerance and improve healthy gut development in recipient preterm infants. The investigators expect to find FFT safe and with fewer cases of NEC and sepsis. The investigators do not expect to prove the effect of the intervention in this study. However, the investigators aim to follow up with a double-blinded multicenter randomized control trial - powered to document our hypothesis - that when colonizing with a healthy microbiome, it is possible decrease incidence of NEC in premature infants.

ELIGIBILITY:
Inclusion criteria for participant preterm infants

* Preterm infants born between GA 26+0 and 30+6
* Delivery at RH or transferred to RH NICU within 24 hours of delivery
* Children administered prophylactic antibiotics due to maternal risk factors, specifically: premature rupture of membranes, groub b streptococcus positive, feber during labour
* Signed parental consent

Exclusion criteria for participant preterm infants

* Major congenital anomalies or birth defects
* Antibiotics for more than 72 hours after birthExtremely SGA infant (weight SD score < -3 SD)
* Need for mechanical ventilation or cardiovascular support before first FFT treatment

Inclusion criteria for mothers of participants

* Women aged 18-45
* Ability to give informed consent

Exclusion criteria for participant mothers

● Mothers who have severe infection, defined by need for other treatment to support infection-related comorbidities, besides from antibiotics (e.g. inotropic treatment, iv fluid resuscitation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
No serious adverse events | 14 days
  No increased incidence of sepsis, NEC and death in the treatment group

SECONDARY OUTCOMES:
Feeding tolerance | 1 month
  Using a standardized clinical scoring system, nurses at our NICU will evaluate any negative reactions to enteral feeding. It includes evaluation of aspirate, feces, amount of enteral nutrition administered, objective evaluation of the abdomen, and signs of obstipation
Microbiota Composition | 1 month
  Total genomic DNA will be subjected to deep metagenome sequencing and related to the study outcomes. When extracting faecal DNA as well as viral DNA/RNA, physical fractionation or selective lysis will be employed to ensure host DNA is kept to a minimum. Remaining host DNA material will be removed during bioinformatics filtering and mapping of the shotgun metagenomics data.
Time to full enteral feeding | 1 month
Blood pressure | 1 month
  Blood pressure in mmHg
Temperature | 1 month
  Rectal temperature in degrees celsius
Pulse | 1 month
  Pulse measured using samsung monitoring equipment according to standard at our NICU
Length | 1 month
  Length in cm
Weight | 1 month
  Weight in kilograms
Stool characteristics - Amount | 1 month
  Score from 1-4 using Amsterdam stool scale
Stool characteristics - Consistency | 1 month
  Score from 1-6 using diapered infant stool scale
Stool characteristics - Color | 1 month
  Score from 1-6 using Amsterdam Stool Scale
Days of hospitalization | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lise Aunsholt, md, phd, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
An anonomized version of the data will be published along with the main report from the intervention study
Supporting Information: Study Protocol, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Kappel SS, Jakobsen GR, Oestergaard KL, Brunse A, Nielsen DS, Aunsholt L. Parental Consent to a Neonatal Clinical Study: The Roles of Uncertainty, Burden of Sample Collection and Societal Expectations. Acta Paediatr. 2025 Oct 6. doi: 10.1111/apa.70333. Online ahead of print. PMID 41051016

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT05272579/Prot_SAP_000.pdf